CLINICAL TRIAL: NCT04993820
Title: The Effects of a Mobile-Application and Text-Message Based Physical Activity Intervention on Physical and Mental Health in People Living With HIV
Brief Title: The Effects of a Mobile-Application Based Physical Activity Intervention in PLWH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Queens College, The City University of New York (Other)
Collaborators: City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-0494
Record Dates: First submitted 2021-06-23; First posted 2021-08-06 (Actual); Last update posted 2021-08-06 (Actual); Status verified 2021-07

CONDITIONS: HIV
Keywords: Physical Activity; RCT
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a physical activity group oran education control group for the the length of the intervention (12 weeks).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Physical Activity (PA) (Experimental): Combination of aerobic exercise and muscle strengthening exercise.
  Interventions: Behavioral: Physical activity
- Education Control (CON) (Active Comparator): No exercise group.
  Interventions: Behavioral: Education control

INTERVENTIONS:
Behavioral: Physical activity — The goal for week one will be to increase moderate-to-vigorous PA (MVPA) by 90 weekly/mins, and by 120 weekly/mins on week two. This amount of time will provide the participant with an adaptation period. The goal for weeks 3-12 will be to increase MVPA by at least 150 weekly/mins. The prescribed aerobic activities can be performed either: 1) outdoors (e.g., walking or cycling), 2) at home (e.g., in-place jogging, dancing, aerobics), or 3) with available exercise equipment if the participant already has this access. Participants will perform a series of 6 to 8 muscle strengthening (MS) exercises for the major muscle groups using elastic bands and their own bodyweight 3 times per week. All MS activities will be depicted in instructional videos available through the app. Participants will be asked to perform 2 sets of 8 to 12 repetitions (reps) per exercise during weeks 1-3, 3 sets of 8 to 12 reps per exercise during weeks 3-7, and 4 sets of 8 to 12 reps per exercise during weeks 8-12.
  Arms: Physical Activity (PA)
Behavioral: Education control — Participants in the education CON group will be asked to perform their usual activities and to not engage in additional PA during the intervention. Participants will receive weekly brochures and reading materials including topics related to living with HIV, healthy eating, stress management, and current Federal PA guidelines for Americans. The brochures and reading materials will be available through the BluejayEngage health web-based platform app.
  Arms: Education Control (CON)

SUMMARY:
A series of adverse physical and mental health effects are often reported among people living with HIV (PLWH) as a consequence of the infection and ART use. Physical activity (PA) has been linked to improved physical an mental health in PLWH. However, Most interventions in the HIV literature evaluating the effects of PA on physical and mental health have included face-to-face supervised exercise in highly controlled environments which is not representative of how the majority of this population engages in PA. Mobile application (app) and text-message based PA interventions are a safe and innovative approach for the delivery of PA programs aimed at improving physical and mental health without the need of direct supervision. Nonetheless, the use of these types of interventions have not been well evaluated in PLWH. Therefore the purpose of this study is to evaluate the effects of a 12-week mobile app and text-based PA intervention on physical and mental health in PLWH.

Participants in the PA group will be given a PA program delivered through a mobile health app which will be accessed through smartphones. As part of the program, weekly text messages will be sent to encourage PA participation. The goal of the intervention is to increase moderate to vigorous PA (MVPA) by at least 150 weekly/mins. The PA program will also include muscle strengthening exercises. Investigators expect improvements in mental health outcomes (i.e., depressive symptoms and HRQoL) and cardiometabolic outcomes (i.e., cardio-autonomic function, body fat percentage, physical activity, and functional exercise capacity) in the PA group when compared to the CON group at the end of 12-weeks.

DETAILED DESCRIPTION:
People living with HIV (PLWH) now live longer due to the effectiveness and availability of anti-retroviral therapy (ART). However, a series of adverse physical and mental health effects are often reported in this population as a consequence of the infection and ART use. Poor mental health and health-related quality of life (HRQoL) is more prevalent among PLWH, with rates of depression as high as 42% and rates of generalized anxiety disorders. recently reported at ~19%. Research also suggests that a number of physical health and cardiometabolic side effects are associated with the disease progression and ART use, and these side effects have led to a significant increase in the risk of cardiovascular disease (CVD) among this patient population .

Among PLWH, physical activity (PA) has been linked with HRQoL , and less anxiety and depression . Furthermore, PA has also been associated with cardiometabolic health benefits , improved body composition , lower diabetes rates , functional exercise capacity , and improved cardio-autonomic function among PLWH, all which can reduce the risk of CVD. However, research suggests that lack of PA combined with sedentary behavior is prevalent among PLWH . A recent meta-analysis showed that PLWH spend approximately 98.6 minutes per day physically active, which is less than the amount reported for other chronic diseases and in general population.This is concerning since physical inactivity is one of the leading risk factors for non-communicable diseases like CVD, diabetes and cancer. Overall these results suggest that PLWH are not engaging in sufficient PA, and thus not receiving the health-related benefits associated with a physically active lifestyle.

Most interventions in the HIV literature evaluating the effects of PA in physical and mental health have included face-to-face supervised exercise in highly controlled environments. However, PA interventions that include supervision in a controlled setting may not be representative of how the majority of PLWH engage in PA. In addition, since the HIV infection is concentrated among those of lower socioeconomic status (SES), access to exercise facilities and regular supervision during PA may be difficult for most PLWH. Recently, investigators conducted a combined home and lab-based aerobic exercise intervention in PLWH and found encouraging results in the adherence rates in the home-based unsupervised sessions (i.e., >80%), suggesting that PLWH will engage in exercise even when there is no direct supervision. To date, a very limited number of studies have evaluated the effectiveness of unsupervised PA interventions in PLWH. Both studies showed that these types of interventions are safe and can be effective at improving physical and mental health outcomes in PLWH.

Mobile application (app) and text-message based PA interventions are a safe and innovative approach for the delivery of PA programs aimed at improving PA participation, reducing sedentary behavior and improving physical and mental health outcomes in a variety of populations, despite the lack of supervision inherent to this design. The use of a mobile app can promote greater engagement as it provides: 1) instructional videos of activities that the participant can safely perform without the need of supervision, 2) an interactive way for participants to track their progress towards meeting the goal volume of weekly PA, and 3) feedback on their PA participation through the integration of text-messaging. The use of text-messaging can be an effective way to provide statements to encourage PA participation, provide counseling on how to overcome barriers to engaging in regular PA and give individualized feedback on current PA participation. In addition, the widespread use of smart phones in the United States, even among those of lower SES, makes these types of interventions an accessible, easy to use and low-cost method to promote PA participation and improve health. However, the use of these types of interventions have not been well evaluated in PLWH. To the best of our knowledge, only one pilot study evaluated the effects of a mobile app exercise intervention in PLWH. Nonetheless, this study lacked a no-exercise control group, included partial supervised and did not include text messaging based on established health behavior models to promote behavior change. The proposed project is innovative as it will be the first randomized controlled trial to test the effects of a mobile app and text-message based PA intervention on physical and mental health outcomes in PLWH. Therefore, the primary aims of this study are:

1. To evaluate the effects of a mobile app and text-based PA intervention on physical health (i.e., HRQoL, perceived physical health, body composition, functional exercise capacity and cardio-autonomic function) in PLWH.

   H1: The mobile app and text-based PA intervention will improve physical health in PLWH at the end of 12 weeks when compared to the education control group.
2. To evaluate the effects of a mobile app and text-based PA intervention on mental health (i.e., depressive symptoms, perceived mental health and health related quality of life) in PLWH.

   H2: The mobile app and text-based PA intervention will improve mental health in PLWH at the end of 12 weeks when compared to the education control group.
3. To evaluate the effects of a mobile app and text-based PA program on PA participation in PLWH.

H3: The mobile app and text-based PA intervention will increase PA participation in PLWH at the end of 12 weeks when compared to the education control group.

Overview and study design The pilot study is a mobile-app and text-message based PA intervention lasting a total of 12-weeks using a randomized controlled design in which adult PLWH (n=40) will be recruited. The study will include two groups: a physical activity (PA) group and an education control (CON) no-exercise group for comparison purposes. Outcome measures will include: perceived physical and mental health, depression symptoms, HRQoL, cardio-autonomic function, body composition, functional exercise capacity and objectively measured PA and sedentary time.

Screening A phone pre-screening will be conducted for all volunteers to explain the purpose and procedures of the study and determine eligibility. Participants will also be asked to bring their most recent (≤ 6 months) CD4 T-cell, HIV viral load and HIV medications to the first lab visit for safety and to determine eligibility.

Baseline Sessions Two baselines sessions will be conducted at the beginning of the study. The baseline sessions will take place seven days apart. During the first session investigators will collect sociodemographic data, evaluate the participant's medical history and HIV status. During the first baseline session investigators will also give the participants a research-grade accelerometer to wear in order to measure their PA and sedentary time for 7-consecutive days. During the second baseline visit investigators will assess the participant's physical health and mental health, depression symptoms, HRQoL, resting heart rate variability (HRV), functional exercise capacity and body composition, and retrieve the accelerometer. The participants will be then randomized to either the PA or CON group. Before the visit participants will be instructed to not consume food, caffeine, tea or tobacco products for at least 3 h before, to refrain from consuming alcohol for at least 48 h before, and to not engage in any exercise for at least 24 h before as this may affect some of the study outcome measures.

Intervention 40 participants will be randomly assigned to either 1) a PA intervention group, or 2) an education CON group (detailed in the intervention section).

Post Intervention Sessions Two post-intervention sessions will be conducted at the end of the study to evaluate changes over time in the main study outcomes. The two sessions will take place 7-days apart. During the first post-intervention session investigators will give the participants an accelerometer to wear in order to measure their PA and sedentary time for 7-consecutive days. During the second visit investigators will assess the participants physical and mental health, depression symptoms, HRQoL, HRV, body composition, functional exercise capacity and retrieve the accelerometers.

ELIGIBILITY:
Inclusion Criteria:

* 1) diagnosed with HIV,
* 2) receiving the same ART for at least six months,
* 3) being clinically stable (i.e., no recent AIDS-defining opportunistic infections, a CD4+ T-cell count ≥ 200 cells·mm-3, and asymptomatic),
* 4) owning a smartphone with text message capabilities, and
* 5) willing to receive four or more text messages per week.

Exclusion Criteria:

* 1) having a diabetes mellitus diagnosis
* 2) requiring the use of an assistive device for walking as it will impair physical activity,
* 3) participating in any sport or planned exercise program on more than two days per week
* 4) having any signs or symptoms of CVD or any known uncontrolled cardiovascular, pulmonary or neuromuscular disease that may preclude exercise participation,
* 5) severe arthritis, hip or knee fracture or spinal surgery in the past 6 months
* 6) having any contraindications to exercise as identified by the American College of Sports Medicine

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Physical Activity (PA) | 7 consecutive days before the start of the intervention and 7 consecutive days during the last week of the intervention
  Minutes of moderate to vigorous PA per week using an Actigraph triaxial accelerometer (Model GT9X) worn at the wrist. This will be done to evaluate for changes in free-living PA as a result of the intervention

SECONDARY OUTCOMES:
Body fat percentage | 12 weeks
  Body fat percentage will be measured through air displacement plethysmography (ADP;BodPod) to evaluate for changes in body composition with the intervention. The ADP will be performed according to manufacturer's guidelines
Fat free mass | 12 weeks
  Fat free mass in kilograms (kg) will be measured through air displacement plethysmography (ADP;BodPod) to evaluate for changes in body composition with the intervention. The ADP will be performed according to manufacturer's guidelines
Cardio-autonomic function | 12 weeks
  Assessed through heart rate variability (HRV) to evaluate for changes in cardio-autonomic function as a result of the intervention. HRV will be measured with the participant in supine position in a dimly lit and quiet environment after 10 minutes of rest. A random 5-minute section of the HRV recording will be utilized for the analysis. A BioRadio (Model BR500) will be utilized to record ECG data through a 1-lead bipolar configuration in order to calculate HRV.
Functional exercise capacity | 12 weeks
  Functional exercise capacity will be measured using the six-minute walk test (6MWT) on a treadmill. The 6MWT test will be performed to evaluate for changes in the estimated maximal oxygen uptake with the intervention following established guidelines.
Depression symptoms | 12 weeks
  Depression symptoms will be measured using the Beck Depression Inventory-II (BDI-II) questionnaire in order to evaluate for changes as a result of the intervention. The instrument includes 21 questions about how the participant has been feeling in the past 2 weeks. BDI-II items are rated on a 4-point scale ranging from 0 to 3 based on severity of each item. The minimum total score is 0 and the maximum total score is 63. The higher the score the worse the severity of depressive symptoms.
Health-related quality of life (HRQoL) | 12 weeks
  HRQoL will be evaluated using the Medical Outcomes Study 36- Item Short-Form Survey (SF-36). The SF-36 includes a total of 36 questions measuring eight different health concepts. The response choices for most items are Likert scales, while Items that assess problems with work or other regular daily activities due to either physical health or emotional problems are dichotomous (yes/no). Each item is scored on a 0 to 100 range with the lowest being a 0 and the highest possible score a 100. Higher scores indicate a more favorable health state. The SF-36 will be used to evaluate for changes in HRQoL as a result of the intervention.
Questions on physical and mental health | 12 weeks
  Overall health status will be assessed through 4 validated short questions from the 2018 BRFSS. The questions ask about the participant's perception of their current general health in a Likert scale, the number of days during the past 30 days their physical health was not good, the number of days during the past 30 days their mental health was not good and number of days in the last 30 days their physical or mental health kept them from doing their usual activities.

CONTACTS AND LOCATIONS:
Overall Officials: Norberto Quiles, Ed.D., Principal Investigator — Queens College of The City University of New York

IPD SHARING:
Plan to Share IPD: No